CLINICAL TRIAL: NCT00127985
Title: The Effect of 6-Methyl-Prednisolone on Organ Dysfunction and Mortality of Patients With Unresolving Multiple Organ Dysfunction Syndrome
Brief Title: 6-Methyl-Prednisolone for Multiple Organ Dysfunction Syndrome
Acronym: NAIF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Principe de Asturias (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Miguel Sanchez Garcia, MD, PhD, Hospital Principe de Asturias
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAIF6MPMODS088UNK9071296
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Multiple Organ Dysfunction Syndrome
Keywords: multiple organ dysfunction syndrome; corticosteroids; mortality
MeSH Terms: conditions — Multiple Organ Failure | interventions — methyl 11,17,21-trihydroxy-3,20-dioxopregna-1,4-diene-16-carboxylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): IV 6-methyl-prednisolone
  Interventions: Drug: 6-methyl-prednisolone
- Comparator (Placebo Comparator): IV Placebo
  Interventions: Drug: 6-methyl-prednisolone

INTERVENTIONS:
Drug: 6-methyl-prednisolone — iv, 2 mg/kg/day, qid

SUMMARY:
Background: Systemic corticosteroids are considered in patients with an adverse clinical course suffering from conditions like the acute respiratory distress syndrome (ARDS) and septic shock. Treated patients not only show improved respiratory function, but also hemodynamic status and overall multiple organ dysfunction score.

Objective: To evaluate the safety and effectiveness of 6-methyl-prednisolone on the clinical course of multiple organ dysfunction syndrome (MODS).

Design: Multi-center, double-blind, randomized, placebo-controlled.

Intervention: Intravenous administration of 6-methyl-prednisolone or placebo (aqueous solution). The duration of the study medication administration protocol is 32 days (1).

Primary Endpoints:

1. All cause Intensive Care Unit (ICU) and 28-day mortality
2. Organ dysfunction score on days 4, 7, 14, and 28 of the protocol.

DETAILED DESCRIPTION:
Background:

Worldwide intensive care physicians consider administering systemic corticosteroids in patients with an adverse clinical course suffering from conditions like the acute respiratory distress syndrome (ARDS) and septic shock. Data from recent small studies performed in patients with unresolving ARDS (1;2) suggest survival benefits associated with rescue therapy with relatively prolonged courses of corticosteroids. Treated patients not only show improved respiratory function, but also hemodynamic status and overall multiple organ dysfunction score. It has been suggested that that the integrity of the hypothalamic-pituitary-adrenal axis may be impaired in this patient subset (3;4)

Objective(s):

To evaluate the safety and effectiveness of a non-selective anti-inflammatory strategy, i.e. 6-methyl-prednisolone, on persistent and unresolving inflammatory states, i.e. multiple organ dysfunction syndrome, on the degree of organ dysfunction and mortality.

Design:

Multi-center, double-blind, randomized, placebo-controlled. Randomization and data entry is internet based (htpp://www.webnaif.com). Patients will be randomized through a computer-generated random-number table and stratified by center in blocs of 6. Sample size, by group 120 patients. The study is powered to detect a 20% reduction in mortality, from 50% to 30% in 100 patients per study group at the 5% significance level with a power of 80%. An additional 20% (n=20) per group have been planned to compensate for losses.

Main Inclusion Criteria:

* Patients with established, unresolving, refractory MODS, in whom all reversible and treatable causes of persistent MODS have been treated or ruled out.
* Patients under endotracheal intubation and mechanical ventilation for at least 7 days.
* Aggregate Multiple Organ Dysfunction Score (5) of greater than 8 over the first seven days of mechanical ventilation and greater than 5 on the day of inclusion.
* Written informed consent to participate in the trial signed by next of kin or other authorized person.

Additional Inclusion Criteria:

* Main cause or disease at admission: Adequate "source control" is required and refers to optimal, complete, and definitive surgical and/or medical therapy.
* Infections:

  1. Infectious causes of persistence of MODS have reasonably been ruled out on clinical or other grounds (infectious endocarditis, undrained abscesses like sinusitis, empyema or abdominal pus). Consider sampling for culture of broncho-alveolar lavage fluid, protected specimen brush or other (empyema fluid, lung tissue) in order to rule out respiratory infection, as well as intra-vascular catheter change and culture.
  2. Present or previous infections, either documented or strongly suspected, have been treated for at least 3 days before inclusion.
* Supportive Care: Optimal hemodynamic, renal, hematologic, nutritional "supportive care" is provided.

Exclusion Criteria:

* Decision not to provide full support.
* Immune status and steroid therapy.

  1. Steroid therapy

     * Currently indicated for chronic or concurrent disease (meningitis, auto-immune disease, asthma, acute exacerbation of COPD, or other). Inhaled steroids are allowed.
     * Administered during current admission (> 20 mg/day of 6-methyl-prednisolone or equivalent for >48 hours).
     * Chronic steroid therapy prior to current admission (> 20 mg of 6-methyl-prednisolone or equivalent/day for > 1 month during previous 3 months).
  2. Other immune-suppressive therapy within the previous 6 months.
  3. Known AIDS.
  4. Neutropenia < 500/mcl.
  5. Preceding organ transplantation.
* Irreversible and or ultimately fatal clinical conditions like metastatic malignant disease or cardiogenic shock caused by coronary artery disease.
* Presence of invasive fungal infection
* Other significant pre-existing underlying chronic diseases:

  1. Severe parenchymal liver disease (Child-Pugh grade C)
  2. Severe and irreversible acute or chronic central nervous system disease.
  3. Severe end-stage chronic obstructive pulmonary disease (home oxygen or more than 1 exacerbation in previous year)
  4. End-stage renal disease (Chronic dialysis).
* Age less than 18 years.
* Pregnancy.
* Morbid obesity: body mass index above 40.
* Recent (last 3 months) upper GI hemorrhage.
* Extensive burns (>30% BSA)
* Known allergy to steroids.
* Written informed consent not available.

Intervention:

Intravenous administration of 6-methyl-prednisolone or placebo(aqueous solution). The duration of the study medication administration protocol is 32 days (1):

* Initial iv loading dose of 160 mg.
* An iv bolus injection of 6-methyl-prednisolone is administered every 6 hours:

  1. 40 mg on days 1 to 14,
  2. 20 mg on days 15 to 21,
  3. 10 mg on days 22 to 28,
  4. 5 mg on days 29 and 30, and
  5. 2.5 mg on days 31 and 32.

Informed consent form and information sheet have been reviewed and approved by the regional Ethics Committee of Madrid (10 centres), the local review boards of the other participating centres, and the Agencia Española del Medicamento (Spanish Ministry of Health).

Ethical Approval:

The study protocol has been approved by the regional Ethics Committee of Madrid (10 centres), the local review boards of the other participating centres, and the Agencia Española del Medicamento (Spanish Ministry of Health).

Stopping Rules:

The independent Data Monitoring Committee (DMC) will have real-time access to the main variable "28-day mortality" (and allocation to study group "A" or "B") and will propose premature interruption of the trial based on sequential analysis if significant differences become apparent. The DMC will perform 5 interim analysis, one every 48 included patients and the criterium used will be a statistically significant difference at the level of p < 0,01 (S.J. Pocock. Clinical Trials. A practical Approach. John Wiley & Sons. New York. 1994).

Primary Endpoints:

1. All cause ICU and 28-day mortality
2. Organ dysfunction score on days 4, 7, 14, and 28 of the protocol.

Planned Subgroup Analysis:

No subgroup analysis are planned.

Side-effects Quantification:

The investigators will use the NIH Toxicity Form with a scale from 1 to 5. Severe adverse events in this severely ill population are precisely defined and require immediate (less than 24 hours) communication to the study website. The DMC will have access to the variables that define and describe the SAEs.

Analysis Plan:

Main comparisons are 28-day and ICU mortality between study groups (chi square test for percentages and log-rank test Kaplan-Meier survival curves. Multiple organ dysfunction score and Sequential Organ Failure Assessment score will be compared at baseline and on days 4, 7, 14 and 28 (Student's t test and/or non-parametric tests). Independent risk factors for mortality will be studied by multivariate analysis (Cox regression) of significant comparisons of the univariate analysis. Analysis sample according to the principle of intention to treat.

Finishing Date:

The finishing date is 18 months after the first inclusion at each centre. Scheduled beginning of the trial is August 2005

Reporting Date:

First trimester 2007.

A large study like the present trial is required to obtain definitive data about safety and effectiveness of 6-methyl-prednisolone administered as rescue therapy in patients with the multiple organ dysfunction syndrome.

Reference List

1. Meduri GU, Headley AS, Golden E, Carson SJ, Umberger RA, Kelso T et al. Effect of prolonged methylprednisolone therapy in unresolving acute respiratory distress syndrome: a randomized controlled trial. JAMA 1998;280(2):159-65.
2. Biffl WL, Moore FA, Moore EE, Haenel JB, McIntyre RC, Jr., Burch JM. Are corticosteroids salvage therapy for refractory acute respiratory distress syndrome? Am.J.Surg. 1995;170(6):591-5.
3. Marik PE, Zaloga GP. Adrenal insufficiency during septic shock. Crit Care Med. 2003;31(1):141-5.
4. Loisa P, Rinne T, Kaukinen S. Adrenocortical function and multiple organ failure in severe sepsis. Acta Anaesthesiol.Scand. 2002;46(2):145-51.
5. Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995;23(10):1638-52.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria:

Patients with established, unresolving, refractory MODS, in whom all reversible and treatable causes of persistent MODS have been treated or ruled out:

* Patients under endotracheal intubation and mechanical ventilation for at least 7 days.
* Aggregate Multiple Organ Dysfunction Score (5) of greater than 8 over the first seven days of mechanical ventilation and greater than 5 on the day of inclusion.
* Written informed consent to participate in the trial signed by next of kin or other authorized person.

Additional Inclusion Criteria:

* Main cause or disease at admission: Adequate "source control" is required and refers to optimal, complete, and definitive surgical and/or medical therapy.
* Infections:

  1. Infectious causes of persistence of MODS have reasonably been ruled out on clinical or other grounds (infectious endocarditis, undrained abscesses like sinusitis, empyema or abdominal pus). Consider sampling for culture of broncho-alveolar lavage fluid, protected specimen brush or other (empyema fluid, lung tissue) in order to rule out respiratory infection, as well as intra-vascular catheter change and culture.
  2. Present or previous infections, either documented or strongly suspected, have been treated for at least 3 days before inclusion.
* Supportive Care: Optimal hemodynamic, renal, hematologic, nutritional "supportive care" is provided.

Exclusion Criteria:

* Decision not to provide full support.
* Immune status and steroid therapy.

  1. Steroid therapy

     * Currently indicated for chronic or concurrent disease (meningitis, auto-immune disease, asthma, acute exacerbation of chronic obstructive pulmonary disease [COPD], or other). Inhaled steroids are allowed.
     * Administered during current admission (> 20 mg/day of 6-methyl-prednisolone or equivalent for >48 hours).
     * Chronic steroid therapy prior to current admission (> 20 mg of 6-methyl-prednisolone or equivalent/day for > 1 month during previous 3 months).
  2. Other immune-suppressive therapy within the previous 6 months.
  3. Known AIDS.
  4. Neutropenia < 500/mcl.
  5. Preceding organ transplantation.
* Irreversible and or ultimately fatal clinical conditions like metastatic malignant disease or cardiogenic shock caused by coronary artery disease.
* Presence of invasive fungal infection
* Other significant pre-existing underlying chronic diseases:

  1. Severe parenchymal liver disease (Child-Pugh grade C)
  2. Severe and irreversible acute or chronic central nervous system disease.
  3. Severe end-stage chronic obstructive pulmonary disease (home oxygen or more than 1 exacerbation in previous year)
  4. End-stage renal disease (Chronic dialysis).
* Age less than 18 years.
* Pregnancy.
* Morbid obesity: body mass index above 40.
* Recent (last 3 months) upper gastrointestinal [GI] hemorrhage.
* Extensive burns (>30% body surface area [BSA])
* Known allergy to steroids.
* Written informed consent not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
All cause ICU and 28-day mortality | 28 days
Organ dysfunction score on days 4, 7, 14, and 28 of the protocol | Days 4, 7, 14, and 28.

SECONDARY OUTCOMES:
Mortality | 28 days
Morbidity: Duration of mechanical ventilation and endotracheal intubation (also a surrogate for acute steroid myopathy) | 28 days
Length of ICU-stay | 28 days
Complications of steroid therapy | 28 days
Infections acquired during the protocol | 28 days
Other complications (hyperglycemia, GI bleeding, acute myopathy, pneumothorax) | 28 days
Adrenal reserve as evaluated by adrenocorticotropic hormone (ACTH) test. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Sanchez, MD, PhD, Study Chair — Hosp. Univ. Principe de Asturias
Locations (6):
- Spain (6):
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Francisco Ortuño Anderiz, Madrid, Madrid
  - Clinica Moncloa, Madrid, Madrid
  - María Mar Cruz Acuaroni, Toledo, Toledo

REFERENCES:
- [Background] Meduri GU, Headley AS, Golden E, Carson SJ, Umberger RA, Kelso T, Tolley EA. Effect of prolonged methylprednisolone therapy in unresolving acute respiratory distress syndrome: a randomized controlled trial. JAMA. 1998 Jul 8;280(2):159-65. doi: 10.1001/jama.280.2.159. PMID 9669790
- [Background] Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995 Oct;23(10):1638-52. doi: 10.1097/00003246-199510000-00007. PMID 7587228